CLINICAL TRIAL: NCT03235908
Title: Copeptin - A Biomarker to Improve Outcome Prediction in Patients With an Acute Psychotic Episode
Brief Title: Copeptin in Outcome Prediction of an Acute Psychotic Episode
Acronym: CoPsych
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-02198
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Acute Psychotic Episode; Schizophrenia Spectrum and Other Psychotic Disorders; Affective Disorder; Bipolar Disorder
Keywords: Copeptin; Outcome prediction
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Mood Disorders; Bipolar Disorder; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Copeptin, Cortisol, Serum Sodium, Urinary sodium and urinary osmolality in case
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an acute psychosis: Acute psychosis in schizophrenia spectrum disorder, affective disorder and bipolar disorder; Observation only
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Observation only

SUMMARY:
An acute psychotic episode is a severe psychiatric syndrome which might occur in different psychiatric diagnoses.

The outcome prediction of relapse rate of a psychotic episode within a certain time frame is difficult and depends on many factors. More and better predictors are required to improve the outcome prediction in order to adjust therapy and follow-up if patients suffer from this acute disease.

Copeptin, a surrogate marker for vasopressin, has been proven helpful in the prediction of the outcome in serious somatic diseases. Additionally, a rise of copeptin due to psychological stress was shown.

The aim of this study is to investigate the association of the neuroendocrine biomarker copeptin and the prediction of the onset of psychotic episode within one year.

DETAILED DESCRIPTION:
An acute psychotic episode is a severe psychiatric syndrome characterised by symptoms like delusions, hallucinations, and perceptual disturbances. A psychotic episode might occur in different psychiatric diagnoses, such as schizophrenia spectrum disorders and affective disorders (depression and bipolar).

The outcome prediction of relapse rate of a psychotic episode within a certain time frame is difficult and depends on many factors. More and better predictors are required to improve the outcome prediction in order to adjust therapy and follow-up if patients suffer from this acute disease.

Copeptin, a surrogate marker for vasopressin, has been proven helpful in the prediction of the outcome in serious somatic diseases such as stroke, myocardial infarction, and pneumonia. Additionally, a rise of copeptin due to psychological stress was shown.

Some studies have shown an increase in vasopressin levels during acute psychosis, no study has been performed using copeptin.

The aim of this study is to investigate the association of the neuroendocrine biomarker copeptin and the prediction of the onset of psychotic episode within one year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Acute psychotic episode
* Informed consent as documented by signature

Exclusion Criteria:

* Limited discernment due to psychiatric disorder to give informed consent
* Acute psychotic Episode due to any organic reason
* Psychotic Episode due to psychotropic substances
* Severe somatic disease (acute myocardial infarction, acute sepsis, acute stroke)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are hospitalized with an acute psychotic episode within schizophrenia spectrum disorder, affective disorder and bipolar disorder.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Copeptin level | One year
  Association of copeptin at inclusion with relapse rate of a psychotic episode within one year

SECONDARY OUTCOMES:
Change in copeptin levels | day 1 until day 30
  Change in copeptin levels from day 1 until day 30
Recovery of psychotic episode | 1 year
  Time until recovery from the Initial psychotic Episode assessed after 30 days and one year
Discharge from hospital | one year
  Time until discharge from hospital assessed after 30 days and one year
Therapy Response assessed by symptom reduction of >30% in PANSS | 30 days
  Therapy Response defined as symptom reduction of >30% in PANSS assessed after 30 days
Therapy Response measured by Global Assessment of Functioning (GAF) scale | 30 days
  Therapy Response measured by Global Assessment of Functioning (GAF) scale assessed after 30 days
Occurence of hyponatremia | 1 day
  Incidence of hyponatremia during an acute psychotic episode assessed at baseline
Occurence of primary polydipsia | 1 day
  Incidence of primary polydipsia in patients with an acute psychotic episode assessed by reported amount of drinking at baseline
number of hospital re-admissions | 1 year
  re-admission rate due to a psychotic episode observed over 1 year
social function after 12 months (functioning) after 12 months assessed by questionnaire | 1 year
  social function after 12 months
Severity of psychotic symptoms after 12 months compared to baseline assessed by questionnaire | 1 year
  Severity of psychotic symptoms (functioning) after 12 months
psychological function (functioning) after 12 months compared to baseline assessed by questionnaire | 1 year
  psychological function (functioning) after 12 months
operational function (functioning) after 12 months compared to baseline assessed by questionnaire | 1 year
  operational function (functioning) after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD-PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schmidt A, Smieskova R, Aston J, Simon A, Allen P, Fusar-Poli P, McGuire PK, Riecher-Rossler A, Stephan KE, Borgwardt S. Brain connectivity abnormalities predating the onset of psychosis: correlation with the effect of medication. JAMA Psychiatry. 2013 Sep;70(9):903-12. doi: 10.1001/jamapsychiatry.2013.117. PMID 23824230
- [Result] Balanescu S, Kopp P, Gaskill MB, Morgenthaler NG, Schindler C, Rutishauser J. Correlation of plasma copeptin and vasopressin concentrations in hypo-, iso-, and hyperosmolar States. J Clin Endocrinol Metab. 2011 Apr;96(4):1046-52. doi: 10.1210/jc.2010-2499. Epub 2011 Feb 2. PMID 21289257
- [Result] Urwyler SA, Schuetz P, Sailer C, Christ-Crain M. Copeptin as a stress marker prior and after a written examination--the CoEXAM study. Stress. 2015 Jan;18(1):134-7. doi: 10.3109/10253890.2014.993966. Epub 2015 Jan 8. PMID 25472823
- [Result] Siegenthaler J, Walti C, Urwyler SA, Schuetz P, Christ-Crain M. Copeptin concentrations during psychological stress: the PsyCo study. Eur J Endocrinol. 2014 Dec;171(6):737-42. doi: 10.1530/EJE-14-0405. Epub 2014 Sep 23. PMID 25249697